CLINICAL TRIAL: NCT04093206
Title: A Double-blind, Randomized, Controlled Study to Compare the Effects of Syrup With EpiCor and Vitamin C to Syrup With Vitamin C Alone on the Common Cold or Influenza in Generally Healthy Children
Brief Title: Compare Effects of EpiCor and Vitamin C to Vitamin C Alone on the Common Cold or Influenza in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Collaborators: Clinres Farmacija d.o.o. (Industry); PharmaLinea d.o.o. (Unknown); Diagnostic Laboratory Medicare PLUS d.o.o. (Unknown); Embria Health Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: EpiCor
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Signs and Symptoms, Respiratory
MeSH Terms: conditions — Signs and Symptoms, Respiratory | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EpiCor and Vitamin C (Experimental): EpiCor (90mg/5ml) and Vitamin C (25mg/5ml) given at dose of 5ml to children 1-2 years old, 7.5ml to children 3-4 years old and 10ml to children 5-6 years old
  Interventions: Dietary Supplement: EpiCor and Vitamin C
- Vitamin C (Active Comparator): Vitamin C (25mg/5ml) given at dose of 5ml to children 1-2 years old, 7.5ml to children 3-4 years old and 10ml to children 5-6 years old
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: EpiCor and Vitamin C — One daily dose
  Arms: EpiCor and Vitamin C
Dietary Supplement: Vitamin C — One daily dose
  Arms: Vitamin C

SUMMARY:
The purpose of the clinical study is to evaluate efficacy of regular daily, 12 weeks, consumption of EpiCor syrup containing EpiCor and vitamin C in non-vaccinated children 1-6 years old on preventing episodes of the common cold and flu as well as on the severity of symptoms of the common cold and flu in case of their occurrence. Additionally, the study aims to assess the effect of EpiCor on the use of prescription drugs and changes of a selected biochemical marker. This is a double-blind, randomized, controlled multi-center clinical trial.

DETAILED DESCRIPTION:
This is a double-blind, randomized, controlled multi-center clinical trial aiming to evaluate the effects of daily consumption of EpiCor with vitamin C, primarily on the incidence and, secondary, on the duration and severity of the common cold and influenza in children, compared to the effects of daily consumption of vitamin C alone. Healthy children aged 1-6 years old are included in the study after parents have provided informed consent for study participation. Children are divided in 3 age groups (1-2 year old, 3-4 years old, 5-6 years old) and randomized in one of the two groups (intervention or control) at a 1:1 ratio. Children eligible for participation are included in the study for 12 weeks. During this period, they visit the investigational center 3 times. During visit 1 (day 0) caregivers get familiarized with the purpose, course and procedures of the trial, provide written informed consent upon which investigator assesses child's suitability for participation and, for eligible children, a study participant number is provided and a randomization number is assigned; in addition, the investigator collects demographic information, data on vital signs, medical history, collects a sample for determination of salivary secretory immunoglobulin A (sIgA), provides caregivers with a Study Dairy and clear instructions regarding completion, consumption, storage and return of unused syrup, taking medication and other food supplements during the study, monitoring adverse events and measures to be taken in the event of serious adverse events, determines the daily dose of syrup to be taken based on child's age, supplies the caregiver with enough syrup and sets a date for next visit. Between visits, children take a prescribed dose of syrup once daily. Six weeks (visit 2) and 12 weeks (visit 3) after the first visit, children and caregivers visit the investigational center again. During these 2 visits, the investigator collects data on vital signs, reviews concomitant medication and the taking of other food supplements, collects sample for determination of salivary SIgA, reviews the Study Dairy, supplies the caregiver with new syrup and provides the same clear instructions as in visit 1. Caregivers are asked to complete the Study Dairy on daily basis and, each time a caregiver marks that a symptom is present, the Investigator receives a notification and reviews the symptoms and consequently confirms the episode of a common cold/flu. The Canadian Acute Respiratory Illness and Flu Scale (CARIFS) is used to assess the severity of symptoms of the common cold and flu in participating children and, in case of occurrence of cold/flu symptoms, caregivers are asked to complete the form twice a day for the first seven days, once on day 10 and once on day 14.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male and female children
* 1-6 years of age
* Children attending kindergarten
* Signed informed consent by child's parent or legal guardian and willingness to participate in all study activities

Exclusion Criteria:

* Immune dysfunction and/or taking an immunosuppressive medication
* Child who has received flu vaccination
* Child who is still breastfed
* Child taking other food supplements
* Unable or unwilling to comply with study protocol, including ingesting investigational product, and completing subject dairy
* Current participation in another clinical study
* Severe co-morbidity or concomitant disease
* Concurrent disease or condition, which in the judgment of the investigator, would make the child inappropriate for participation in the study
* High risk of complications from influenza
* Allergies to yeast-derived products
* Severe environmental allergies requiring medication or need for allergy shots

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Incidence of the common cold an influenza | Number of episodes of common cold and/or influenza during 12 weeks of product consumption
  Daily Study Dairy

SECONDARY OUTCOMES:
Duration of the common cold and influenza | Duration of common cold and influenza during 12 weeks of product consumption
  Daily Study Dairy
Severity of common cold and influenza | Severity of common cold and influenza symptoms during the 12 weeks of product consumption
  Canadian Acute Respiratory Illness and Flu Scale questionnaire
Use of prescription drugs | Number of prescription drugs during the 12 weeks of product consumption
  Daily Study Dairy
Change of salivary secretory immunoglobulin A (sIgA) levels | Change of salivary sIgA levels after 6 and 12 weeks of product consumption
  Salivary sIgA
Safety of investigational product consumption | Safety of investigational product consumption during the 12 weeks study period
  Adverse Events during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Alojz Ihan, Principal Investigator — University of Ljubljana
Locations (21):
- Slovenia (21):
  - Zdravstveni dom Domzale, Domžale
  - Zasebna pediatricna ordinacija Ivan Kauzlaric, Ilirska Bistrica
  - ZD Ivancna Gorica, Ivančna Gorica
  - Zdravstveni dom Kocevje, Kočevje
  - Ambulanta za otroke in solarje Pedenjped d.o.o., Lenart v Slov. Goricah
  - Zasebna ambulanta Moj pediater Matjaz Homsak, Lenart v Slov. Goricah
  - Zasebna otroska in solska ambulanta Mojca Ivankovic Kacjan, Lenart v Slov. Goricah
  - Clinres Farmacija d.o.o., Ljubljana
  - Zdravstveni dom Ljubljana, Ljubljana
  - Zasebna pediatricna ambulanta Vesna Lazar Daneu, Lucija
  - Pediatrinja Suzana Skorjanc Antolic Zdravstvena Dejavnost d.o.o., Maribor
  - Zdravstveni dom Dr. Adolfa Droca Maribor, Maribor
  - Zdravstveni dom Dr. Adolfa Drolca Maribor, Maribor
  - Zasebna pediatricna ambulanta Damir Dabranin, Slovenske Konjice
  - Zdravstveni dom Nova Gorica, Šempeter pri Gorici
  - Pediatrija Sentilj, Šentilj v Slovenskih goricah
  - Zdravstveni dom Tolmin, Tolmin
  - Zadravstveni dom Trebnje, Trebnje
  - Zdravstveni dom Trebnje, Trebnje
  - Zasebna Otroska in Solska Ordinacija, Tržič
  - Zdravstveni dom Zagorje, Zagorje ob Savi